CLINICAL TRIAL: NCT00028483
Title: A Phase II Study Using SGN-15 (cBR96 - Doxorubicin Immunoconjugate) in Combination With Taxotere for the Treatment of Metastatic or Recurrent Breast Carcinoma
Brief Title: Monoclonal Antibody Therapy and Docetaxel in Treating Women With Metastatic or Recurrent Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Purpose: Treatment
Other Study IDs: CDR0000069079; SGEN-UAB-9912; UAB-9912
Record Dates: First submitted 2002-01-04; First posted 2003-06-27 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BR96-doxorubicin immunoconjugate; Docetaxel

INTERVENTIONS:
Drug: cBR96-doxorubicin immunoconjugate
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining docetaxel and monoclonal antibody therapy in treating women who have metastatic or recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and safety profile of doxorubicin-monoclonal antibody BR96 immunoconjugate (SGN-15) and docetaxel in women with metastatic or recurrent breast cancer.
* Determine the clinical response rate and duration of response of patients treated with this regimen.

OUTLINE: Patients receive doxorubicin-monoclonal antibody BR96 immunoconjugate (SGN-15) IV over 2 hours and docetaxel IV over 30 minutes on day 1 of weeks 1-6. Treatment repeats every 8 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A maximum of 45 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or recurrent breast carcinoma

  * Unresectable disease
  * Previously treated with no more than 2 chemotherapy regimens for metastatic disease OR
  * Recurrent within 6 months of adjuvant chemotherapy
* Must have one of the following:

  * Measurable disease
  * Positive bone scan and elevation of serum tumor marker for adenocarcinoma

    * Serum levels must have increased over 2 consecutive measurements and exceed at least 2 times upper limit of normal
* Lewis-y antigen expression documented by immunohistochemistry
* No brain metastases that are uncontrolled or require active treatment (including steroids)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin at least 10 g/dL
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding diathesis

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2.5 times normal
* Alkaline phosphatase no greater than 2.5 times normal (unless documented bony metastasis present)
* Amylase/lipase less than 1.5 times normal
* Hepatitis B and C negative
* No hepatic failure

Renal:

* Creatinine no greater than 1.5 times upper limit of normal
* No renal failure

Cardiovascular:

* LVEF greater than 50% by echocardiogram or MUGA scan
* No congestive heart failure

Other:

* HIV negative
* No antibody present that detects monoclonal antibody BR96 in serum
* No peripheral neuropathy grade 2 or greater
* No dementia or altered mental status
* No other serious underlying medical condition that would preclude study participation
* No prior allergic reactions to recombinant human or murine proteins
* No uncontrolled peptic ulcer disease
* No active viral, bacterial, or systemic fungal infections
* No other primary malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No serious nonmalignant disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 8 weeks since prior therapeutic or diagnostic murine/humanized/human chimeric antibodies

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, carboplatin, mitomycin, or anthracyclines)
* No prior cumulative anthracycline of 300 mg/m2 or more
* No concurrent antineoplastic agents

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior hormonal therapy
* No concurrent hormonal therapy except estrogen replacement

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No other concurrent experimental agents
* No concurrent immunosuppressive medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisle M. Nabell, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States